CLINICAL TRIAL: NCT01572662
Title: Phase II Study of Timed Sequential Busulfan in Combination With Fludarabine in Allogeneic Stem Cell Transplantation
Brief Title: Allogeneic Transplantation Using Timed Sequential Busulfan and Fludarabine Conditioning
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2011-0958; NCI-2012-00573 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2012-04-04; First posted 2012-04-06 (Estimated); Results first posted 2023-06-29 (Actual); Last update posted 2023-06-29 (Actual); Status verified 2023-06

CONDITIONS: Leukemia; Acute Myeloid Leukemia; Acute Lymphocytic Leukemia; Chronic Myeloid Leukemia; Chronic Lymphocytic Leukemia; Myeloproliferative Diseases; Non-Hodgkins Lymphoma; Hodgkins Lymphoma; Multiple Myeloma; Myelodysplastic Syndrome
Keywords: Leukemia; Acute myeloid leukemia; Acute lymphocytic leukemia; Chronic myeloid leukemia; Chronic lymphocytic leukemia; Myeloproliferative Diseases; Non-Hodgkins Lymphoma; Hodgkins lymphoma; Multiple myeloma; Myelodysplastic syndrome; MDS; Fludarabine monophosphate; Fludarabine phosphate; Fludara; Busulfan; Busulfex; Myleran; Tacrolimus; Prograf; Methotrexate; G-CSF; Filgrastim; Neupogen; Stem cell transplant; Allogeneic Transplantation
MeSH Terms: conditions — Leukemia; Leukemia, Myeloid, Acute; Precursor Cell Lymphoblastic Leukemia-Lymphoma; Leukemia, Myelogenous, Chronic, BCR-ABL Positive; Leukemia, Lymphocytic, Chronic, B-Cell; Lymphoma, Non-Hodgkin; Hodgkin Disease; Multiple Myeloma; Myelodysplastic Syndromes | interventions — fludarabine phosphate; Busulfan; Tacrolimus; Methotrexate; Granulocyte Colony-Stimulating Factor; Filgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Fludarabine + Busulfan (Experimental): Fludarabine administered by vein at dose of 40 mg/m2 in 100 ml of normal saline (NS) on Days -6 through -3.
  First two doses of Busulfan, 80 mg/m2 administered as an outpatient or as an inpatient to facilitate for this pharmacokinetically directed therapy. Busulfan is administered at the dose calculated to achieve a total (including first two doses delivered on day -13 and -12) systemic exposure of 20,000 ± 12% µMol-min based on the pharmacokinetic studies.
  Interventions: Drug: Fludarabine monophosphate; Drug: Busulfan; Procedure: Stem Cell Infusion; Drug: Tacrolimus; Drug: Methotrexate; Drug: G-CSF

INTERVENTIONS:
Drug: Fludarabine monophosphate — 40 mg/m2 by vein on Days -6 through -3.
  Other Names: Fludarabine Phosphate; Fludara
Drug: Busulfan — First two doses of Busulfan, 80 mg/m2 administered as an outpatient or as an inpatient to facilitate for this pharmacokinetically directed therapy. Busulfan is administered at the dose calculated to achieve a total (including first two doses delivered on day -13 and -12) systemic exposure of 20,000 ± 12% µMol-min based on the pharmacokinetic studies.
  Other Names: Busulfex; Myleran
Procedure: Stem Cell Infusion — Fresh or cryopreserved bone marrow or peripheral blood progenitor cells infused on Day 0.
Drug: Tacrolimus — Starting dose of 0.015 mg/kg (ideal body weight) as 24 hour continuous infusion daily adjusted to achieve therapeutic level of 5-15 ng/ml. Tacrolimus changed to oral dosing when tolerated and can be tapered off after day +90 if no graft versus host disease (GVHD) present.
  Other Names: Prograf
Drug: Methotrexate — 5 mg/m2 by vein on Days 1, 3, 6 and 11 post transplant.
Drug: G-CSF — 5 mcg/kg/day subcutaneously beginning on Day +7, and continuing until absolute neutrophil count (ANC) is > 500 * 10/L for 3 consecutive days.
  Other Names: Filgrastim; Neupogen

SUMMARY:
The goal of this clinical research study is to learn if giving busulfan and fludarabine before a stem cell transplant can help control the disease better than the standard method in patients with leukemia, lymphoma, multiple myeloma, MDS, or MPD. In this study, 2 doses of busulfan will be given 2 weeks before a stem cell transplant followed by 4 doses of busulfan and fludarabine during the week before the stem cell transplant, rather than the standard method of giving 4 doses of busulfan and fludarabine only during the week before the stem cell transplant.

The safety of this combination therapy will also be studied.

Busulfan is designed to kill cancer cells by binding to DNA (the genetic material of cells), which may cause cancer cells to die. Busulfan is commonly used in stem cell transplants.

Fludarabine is designed to interfere with the DNA of cancer cells, which may cause the cancer cells to die.

DETAILED DESCRIPTION:
Central Venous Catheter:

If you choose to take part in this study, the chemotherapy, some of the other drugs in this study, and the stem cell transplant will be given by vein through your central venous catheter (CVC). A CVC is a sterile flexible tube and needle that will be placed into a large vein while you are under local anesthesia. Blood samples will also be drawn through your CVC. The CVC will remain in your body during treatment. Your doctor will explain this procedure to you in more detail, and you will be required to sign a separate consent form.

Study Drug Administration and Procedures:

For a stem cell transplant, the days before you receive your stem cells are called minus days. The day you receive the stem cells is called Day 0. The days after you receive the stem cells are called plus days.

You will receive a dose of busulfan by vein over about 3 hours on Day -13 and Day -12. With the Day -13 busulfan infusion, about 11 samples of blood (about 1-2 teaspoons each time) will be drawn for pharmacokinetic (PK) testing at various time points before and after you receive your first dose of busulfan. The study staff will tell you the blood testing schedule. PK testing measures the amount of study drug in the body at different time points. The PK testing will help the doctor decide your dose of busulfan for Days -6 through -3. If needed, PK blood testing may also be done on Day -6 during your dose of Busulfan. You may receive the Day -13 and Day -12 busulfan dose either as an outpatient in the clinic or as an inpatient in the hospital.

A heparin lock line will be placed in your vein to lower the number of needle sticks needed for these draws. If it is not possible for the PK tests to be performed for technical reasons, you will be taken off study and receive the standard fixed dose of busulfan.

On Days -13 and -12, you will receive busulfan by vein over 3 hours.

On Days -11 through -7, you will rest.

On Days -6 through -3, you will receive fludarabine by vein over 1 hour, then busulfan by vein over 3 hours.

On Days -2 and -1, you will rest.

On Day 0, you will receive the stem cell transplant by vein.

After the transplant, you will receive tacrolimus, methotrexate, or other drugs to weaken the immune system in the standard manner to lower the risk of graft-vs-host disease (GVHD), a reaction of the donor's immune cells against the recipient's body.

You will receive tacrolimus by vein as a nonstop infusion until you are able to take it by mouth to help lower the risk of GVHD. You will then take tacrolimus by mouth 2 times a day for about 3 months. After that, your tacrolimus dose may be lowered if you do not have GVHD. Your doctor will discuss this with you. On Days 1, 3, and 6, if your stem cells are from a related or matched unrelated donor, you will receive methotrexate over 30 minutes each day by vein to help lower the risk of GVHD. Participants receiving a matched unrelated donor will also receive methotrexate on Day 11 after the transplant.

You will receive filgrastim as an injection under the skin 1 time a day, starting 1 week after the transplant, until your blood cell levels return to normal. Filgrastim is designed to help with the growth of white blood cells.

Study Testing:

While you are in the hospital, you will be checked for any side effects as part of your standard of care. Blood (about 2 teaspoons) will be drawn every day to check for side effects, for routine tests, to check your blood counts, kidney and liver function, and to check for infections.

As part of standard care, you will remain in the hospital for about 3-4 weeks after the transplant. After you are sent home from the hospital, you must remain in the Houston area to be checked for infections and other transplant side effects until about 3 months after transplant. During this time, you will return to the clinic at least 1 time each week. The following tests and procedures will be performed:

* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 2 teaspoons) will be drawn for routine tests.

About 1, 3, 6, and 12 months after the transplant:

* You will have a physical exam, including measurement of your vital signs (blood pressure, heart rate, temperature, and breathing rate).
* You will be asked about how you are feeling and about any side effects you may be having.
* Blood (about 5 teaspoons) will be drawn to see how well the transplant has "taken."
* You will have a bone marrow aspiration to check the status of the disease, if your doctor thinks it is needed. To collect a bone marrow aspiration, an area of the hip or other site is numbed with anesthetic, and a small amount of bone marrow is withdrawn through a large needle.

Length of Study:

You will be taken off study 3 years after the end of treatment. You may be taken off study early if the disease gets worse, if you have any intolerable side effects, of if you are unable to follow study directions.

You should talk to the study doctor if you want to leave the study early. If you are taken off study early, you still may need to return for routine follow-up visits after the transplant, if your transplant doctor decides it is needed.

It may be life-threatening to leave the study after you have begun to receive the study drugs but before you receive the stem cells.

This is an investigational study. Busulfan and fludarabine are both FDA approved and commercially available. The investigational part of this study is the addition of 2 more doses of busulfan.

Up to 200 patients will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with high-risk hematologic malignancies with anticipated poor prognosis with non transplant therapy, including those in remission or with induction failure and after treated or untreated relapse. Diagnoses to be included a) Acute myeloid leukemia; b) Acute lymphocytic leukemia; c) Chronic myeloid leukemia; d) Chronic lymphocytic leukemia; e) Myelodysplastic syndrome; f) Myeloproliferative syndromes; g) Non-Hodgkins lymphoma; h) Hodgkins Lymphoma; i) Multiple myeloma.
2. Patients must have a histocompatible stem cell donor. An HLA-identical related donor or a 8/8 matched unrelated donor.
3. Age 5 to 75 years old.
4. Performance score of >/= 70 by Karnofsky/Lansky or PS 0 to 1 (ECOG </=1).
5. Left ventricular ejection fraction at least 40%.
6. Adequate pulmonary function with FEV1, FVC and DLCO >/=50% of expected corrected for hemoglobin and/or volume. Children unable to perform pulmonary function tests (e.g., less than 7 years old) pulse oximetry of >/= 92% on room air
7. Creatinine clearance (calculated creatinine clearance is permitted) should be >40 ml/min.
8. Bilirubin </= 2 x the upper limit of normal (except Gilbert's Syndrome). SGPT (ALT) < 200.
9. Negative Beta HCG test in a woman with child bearing potential, defined as not post-menopausal for 12 months or no previous surgical sterilization. Women of child bearing potential must be willing to use an effective contraceptive measure while on study.
10. Patient or patient's legal representative, parent(s) or guardian able to sign informed consent.

Exclusion Criteria:

1. HIV seropositivity.
2. Uncontrolled infections.

Ages: 5 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 201 (Actual)
Dates: Start 2012-04-11 (Actual); Primary Completion 2022-08-11 (Actual); Study Completion 2022-08-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Uday Popat, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Popat UR, Mehta RS, Bassett R, Chen J, Valdez BC, Kawedia J, Ahmed S, Alousi AM, Anderlini P, Al-Atrash G, Bashir Q, Ciurea SO, Hosing CM, Im JS, Jones R, Kebriaei P, Khouri I, Marin D, Nieto Y, Olson A, Oran B, Parmar S, Rezvani K, Qazilbash MH, Shah N, Srour SA, Shpall EJ, Champlin RE, Andersson BS. Fludarabine with a higher versus lower dose of myeloablative timed-sequential busulfan in older patients and patients with comorbidities: an open-label, non-stratified, randomised phase 2 trial. Lancet Haematol. 2018 Nov;5(11):e532-e542. doi: 10.1016/S2352-3026(18)30156-X. PMID 30389035
- See also: MD Anderson Cancer Center — http://www.mdanderson.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited from April 2012 to December 2015 at MD Anderson Cancer Center.
Groups:
- Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l; Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.: Allogeneic stem cell transplant for patients with hematologic malignancies: The randomization was stratified equally for the first 100 patients at study entry and conditioned regimen with Fludarabine/Timed Sequential (TS) Busulfan AUC 16,000umol/l vs. Fludarabine/Timed sequential Busulfan AUC 20,000umol/l.
Period: Overall Study
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.
Started | 50 | 151
Completed | 49 | 150
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 0
Not completed — Physician Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l; Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.: Allogeneic stem cell transplant for patients with hematologic malignancies: The randomization was stratified equally for the first 100 patients at study entry and conditioned regimen with Fludarabine/Timed sequential Busulfan AUC 16,000umol/l vs. Fludarabine/Timed Sequential (TS) Busulfan AUC 20,000umol/l.
- Total: Total of all reporting groups
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l. | Total
Number analyzed (Participants) | 49 | 150 | 199
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 1 | 0 | 1
  Between 18 and 65 years | 37 | 94 | 131
  >=65 years | 11 | 56 | 67
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 59 | 72
  Male | 36 | 91 | 127
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 4 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 8 | 10
  White | 44 | 138 | 182
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 49 | 149 | 198
  Saudi Arabia | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Non-Relapse Mortality Rate (NRM)
Description: Number of participants expired within the first 100 days after transplant not due to relapsed disease.
Time Frame: 100 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.
Number analyzed (Participants) | 49 | 150
Participants | 2 | 8

2. Secondary Outcome: Overall Survival
Description: Number of participants that are disease free and alive one year post transplant.
Time Frame: Up to 1 year post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.
Number analyzed (Participants) | 49 | 150
Participants | 29 | 93

3. Secondary Outcome: Overall Survival
Description: Number of participants that were diseased free and alive 3 years post-transplant.
Time Frame: Up to 3 years post-transplant
Measure: Count of Participants; unit: Participants
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.
Number analyzed (Participants) | 49 | 150
Participants | 16 | 47

ADVERSE EVENTS:
Time Frame: Adverse events were collected up to 3 years post transplant.
Arm/Group | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l.
All-Cause Mortality (participants affected / at risk) | 31/49 | 93/150
Serious Adverse Events (participants affected / at risk) | 6/49 | 8/150
Other Adverse Events (participants affected / at risk) | 43/49 | 141/150
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l (N=49) | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l. (N=150)
Skin GvHD (Skin and subcutaneous tissue disorders) | 2 | 6
Bacterial Infections (Infections and infestations) | 6 | 8
Viral Infections (Infections and infestations) | 2 | 4
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 1 | 6
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Transcient Secondary graft failure (Blood and lymphatic system disorders) | 1 | 3
Delayed engraftment (Blood and lymphatic system disorders) | 1 | 0
Primary graft failure (Blood and lymphatic system disorders) | 1 | 0
ABO incompatibility (Blood and lymphatic system disorders) | 2 | 2
Low Platelet (Investigations) | 1 | 0
GI GvHD (Gastrointestinal disorders) | 6 | 5
Liver GvHD (Hepatobiliary disorders) | 3 | 5
Fungal Infections (Infections and infestations) | 0 | 1
Parasite Infections (Infections and infestations) | 0 | 1
Sepsis like syndrome (General disorders) | 0 | 2
HSCT related microangiopathy (TA-TMA) (Blood and lymphatic system disorders) | 0 | 1
Oral mucositis (Gastrointestinal disorders) | 0 | 1
Polyneuropathy (Musculoskeletal and connective tissue disorders) | 0 | 1
Elevated bilirubin (Hepatobiliary disorders) | 0 | 2
VOD/SOS (Hepatobiliary disorders) | 0 | 3
Chronic lung GvHD (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Diverticulitis/neutropenic colitis (Gastrointestinal disorders) | 0 | 1
Autoimmune hemolytic anemia (Immune system disorders) | 1 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm 1: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 16,000 Umol/l (N=49) | Arm 2: Participants w/Hematologic Malignancies Treated w/Fludarabine/TS Busulfan AUC 20,000umol/l. (N=150)
Bacterial Infections (Infections and infestations) | 22 | 82
Parasite Infections (Infections and infestations) | 1 | 0
Fungal Infections (Infections and infestations) | 3 | 8
Viral Infections (Infections and infestations) | 23 | 75
Fevers (General disorders) | 2 | 4
Flu like syndrome (General disorders) | 1 | 0
Fluid overload (General disorders) | 25 | 81
ABO incompatibility (Investigations) | 2 | 0
GI GvHD (Gastrointestinal disorders) | 9 | 37
Liver GvGHD (Investigations) | 10 | 38
Mucositis (Gastrointestinal disorders) | 37 | 141
Upper GI GvHD (Gastrointestinal disorders) | 11 | 34
Liver GvHD (Hepatobiliary disorders) | 6 | 38
Chronic GI GvHD (Metabolism and nutrition disorders) | 1 | 0
Chronic ocular GvHD (Eye disorders) | 10 | 25
Chronic oral GvHD (Gastrointestinal disorders) | 5 | 25
Chronic lung GvGHD (Respiratory, thoracic and mediastinal disorders) | 4 | 9
Neutropenic fevers (Blood and lymphatic system disorders) | 8 | 41
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 7 | 28
Skin GvHD (Skin and subcutaneous tissue disorders) | 29 | 0
Hypertension (Vascular disorders) | 11 | 51
Diarrhea (Gastrointestinal disorders) | 7 | 30
Nausea (Gastrointestinal disorders) | 43 | 119
Hemorrhagic cystitis (Renal and urinary disorders) | 2 | 1
BK virus assoiated Hemorrhagic cystitis (Infections and infestations) | 2 | 20
Elevated transminitis (Investigations) | 22 | 42
Elevated bilirubin (Investigations) | 16 | 57
Encephalopathy (Psychiatric disorders) | 4 | 1
Rash (Skin and subcutaneous tissue disorders) | 4 | 19
Ejection fraction decreased (Cardiac disorders) | 1 | 0
Renal insufficiency (Renal and urinary disorders) | 25 | 25
Chronic Skin GvHD (Skin and subcutaneous tissue disorders) | 3 | 3
Chronic GvHD (Musculoskeletal and connective tissue disorders) | 3 | 3
Chronic vaginal GvHD (Reproductive system and breast disorders) | 3 | 3
Chronic GvHD_Serositis (Respiratory, thoracic and mediastinal disorders) | 2 | 2
BOOP (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Dysrhythmia (Cardiac disorders) | 5 | 5
Ejection fraction decreased (Cardiac disorders) | 4 | 4
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Ascites (Gastrointestinal disorders) | 1 | 1
Diverticulits/colitis (Gastrointestinal disorders) | 2 | 2
PRES (Nervous system disorders) | 4 | 4
Confusions (Psychiatric disorders) | 2 | 2
Hallucination (Psychiatric disorders) | 1 | 1
Headache (Nervous system disorders) | 5 | 5
Tremor (Nervous system disorders) | 2 | 2
Palmar-plantar erythrodysesthesia (Skin and subcutaneous tissue disorders) | 1 | 1
VOD/SOS (Hepatobiliary disorders) | 2 | 2
Autoimmune hemolytic anemia (Investigations) | 4 | 4
Red cell dysplasia due to major ABO incompatibility (Investigations) | 3 | 3
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 2
Thromboembolic event (Vascular disorders) | 1 | 1
Idiopathic thrombocytopenic purpura (ITP) (Investigations) | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-08-02): https://cdn.clinicaltrials.gov/large-docs/62/NCT01572662/Prot_SAP_000.pdf